CLINICAL TRIAL: NCT03286634
Title: Asia-wide, Multicenter Open-label, Phase II Non-randomised Study Involving Children With Down Syndrome Under 21 Year-old With Newly Diagnosed, Treatment naïve Acute Lymphoblastic Leukemia
Brief Title: ASIA Down Syndrome Acute Lymphoblastic Leukemia 2016
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Hospital Organization Nagoya Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASIA-DS-ALL-2016
Record Dates: First submitted 2017-08-09; First posted 2017-09-18 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Down Syndrome; Acute Lymphoblastic Leukemia; Childhood Cancer
MeSH Terms: conditions — Down Syndrome; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms | interventions — Daunorubicin; Prednisolone; prednylidene; Vincristine; Epirubicin; Mercaptopurine; Methotrexate; Hydrocortisone; Cytarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: risk stratification-directed chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SR (Experimental): Standard Risk (SR) :
  CNS 3 or CNS 2 regardless of response OR Time-point #1 (Day 15 induction) Flow MRD ≥ 1% (treatment will not be de-escalated even MRD <0.01% by TP#2) OR Time-point #2 (Day 1 IDMTX/MP of Consolidation) ≥0.01%
  SR strategy:
  All SR patient will have to receive two doses of anthracycline and 12 L-asparaginase doses during induction except those who are escalated to SR at time point 2 when MRD ≥0.01%.
  During the first year of maintenance phase (48 weeks; 4x12 weeks blocks), cyclophosphamide and cytarabine bolus will be administered at 4 weekly interval.
  Interventions: Drug: Daunorubicin; Drug: Prednisolone; Drug: Vincristine; Drug: Epirubicin; Drug: E-coli L-asparaginase; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Hydrocortisone; Drug: Cytarabine; Drug: Cyclophosphamide
- LR (Experimental): Low Risk (LR):
  Time-point #1 (Day 15 induction) Flow MRD <1% AND Time-point #2 (Day 1 IDMTX/MP of Consolidation) <0.01% AND CNS 1 only
  LR strategy:
  For LR patients, one dose of anthracycline and 3 doses of L-asparaginase will be omitted during induction.
  Following re-induction I, interim maintenance and additional block of re-induction ie. re-induction II prior to maintenance phase will be omitted for LR patients.
  Interventions: Drug: Daunorubicin; Drug: Prednisolone; Drug: Vincristine; Drug: Epirubicin; Drug: E-coli L-asparaginase; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Daunorubicin — Given IV
  Other Names: DNR
Drug: Prednisolone — Given PO or IV
  Other Names: Pred
Drug: Vincristine — Given IV
  Other Names: VCR
Drug: Epirubicin — Given IV
  Other Names: EPI
Drug: E-coli L-asparaginase — Given IM or IV
  Other Names: E-coli L-Asp
Drug: 6-Mercaptopurine — Given PO
  Other Names: 6-MP
Drug: Methotrexate — Given IV, PO or IT
  Other Names: MTX
Drug: Hydrocortisone — Given IT
Drug: Cytarabine — Given IV, IT or SC
  Other Names: Ara-C
  Arms: SR
Drug: Cyclophosphamide — Given IV
  Other Names: Cy
  Arms: SR

SUMMARY:
To evaluate the outcome of a prednisolone and low dose methotrexate based protocol in Down syndrome children with ALL (DS-ALL) in an Asia-wide study. The treatment protocol was modified based upon backbone of Taiwan Pediatric Oncology Group (TPOG)-ALL protocol in which risk classification will be guided by level of flow minimal residual disease (MRD) instead.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome diagnosed clinically or cytogenetically (including Mosaic Down)
* Newly diagnosed ALL according to WHO 2016 classification.
* Age < 21 years old at time of enrollment.
* ECOG performance status (PS) score of 0-2.
* Written informed consent obtained from legally acceptable representatives.

Exclusion Criteria:

* Second malignancy.
* Philadelphia positive ALL.
* Mature B-ALL.
* Mixed phenotype acute leukemia.
* Any previous treatment with cytotoxic chemotherapy excluding treatment for TAM or radiation therapy. Patient pre-treated with short term steroid (< 7 days of duration within last 1 month prior to treatment start) can be enrolled into this study.
* Renal dysfunction with creatinine >2x upper limit of normal (ULN). Patients whose creatinine has improved to <2x ULN before treatment commencement can enrol subject to discretion of site PI.
* Liver dysfunction with direct bilirubin > 5x ULN.
* Any serious uncontrolled medical condition or impending end organ dysfunction that would impair the ability of the subject to receive protocol therapy, including:

  1. History of coronary arterial disease, cardiomyopathy, heart failure, arrhythmia (other than sinus arrhythmia) or severe cardiac malformation which with residual abnormalities or requires further major corrective surgery within 2 years.
  2. Ongoing uncontrolled hypertension.
  3. Ongoing uncontrolled diabetes mellitus.
  4. Ongoing uncontrolled infection.
  5. History of congenital or acquired immunodeficiency including HIV infection.
  6. History of interstitial pneumonia, pulmonary fibrosis, bronchiectasis or severe pulmonary emphysema.
  7. CNS hemorrhage.
  8. Psychiatric disorder.
  9. Other concurrent active neoplasms.
* Pregnant or lactating women.
* Doubtful compliance or ability to complete study therapy due to financial, social, familial or geographic reason, or in the judgement of site investigator.

Ages: 0 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-18 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2033-03-31 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | Up to 5 years
  Percentage of patients who are event free at 5 years.

SECONDARY OUTCOMES:
Overall survival | Up to 5 years
  Percentage of patients who survive at 5 years.
Disease free survival | Up to 5 years
  Percentage of patients who are leukemia free at 5 years.
Induction failure | 5 weeks
  Percentage of patients who had failed induction.
Complete remission rate | 5 weeks
  Percentage of patients who had achieved complete remission at the end of induction.
Cumulative incidence of relapse | Up to 5 years
Incidence of treatment-related adverse events | Up to 10 years
  Incidence of treatment-related infectious and metabolic complications (throughout various phases of study therapy) and secondary neoplasms.
Flow MRD at day 15 | At day 15 of induction therapy
  To assess the prognostic value flow MRD level during induction for DS-ALL.

CONTACTS AND LOCATIONS:
Overall Officials: Allen Yeoh, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (10):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Kagoshima University Hospital, Kagoshima, Japan
- Malaysia (2):
  - University of Malaya Medical Centre, Kuala Lumpur
  - Subang Jaya Medical Centre, Subang Jaya
- Singapore (2):
  - National University Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore
- Taiwan (3):
  - National Taiwan University Children's Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Memorial Hopsital, Linkou, Taoyuan District
- Siriraj Hospital Mahidol University, Bangkok, Thailand